CLINICAL TRIAL: NCT00165828
Title: Randomized Trial to Assess Efficacy and Safety of an add-on Treatment With Zonisamide in Adults With Focal Epileptic Seizures With or Without Secondary Generalization
Brief Title: Efficacy and Safety of an add-on Treatment With Zonisamide in Adults With Focal Epileptic Seizures With or Without Secondary Generalization
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai GmbH (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZNS-D-04-001; 2005-000260-57 (EudraCT Number)
Record Dates: First submitted 2005-09-13; First posted 2005-09-14 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2013-11

CONDITIONS: Epilepsy
Keywords: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Zonisamide

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Zonegran
- 2 (Experimental)
  Interventions: Drug: Zonegran

INTERVENTIONS:
Drug: Zonegran — Intravenous injection; initial daily dose of 50 mg zonisamide (2x25 mg) in both treatment groups; following a prospective or retrospective baseline phase of 8 weeks the study drug will be administered twice daily during 16 consecutive weeks.

SUMMARY:
Patients with focal epileptic seizures with or without generalization who are at present treated with one or two antiepileptic drugs are eligible for this study, provided that they fulfill all inclusion criteria and none of the exclusion criteria. Following a baseline phase of 8 weeks duration, the patients are randomised and they receive an initial daily dose of 50 mg zonisamide during the first week. The daily dose is then increased to 200 mg zonisamide in group A or 400 mg zonisamide in group B, respectively. After eight weeks of treatment, the daily dose in group A can be increased to 300 mg in case of insufficient efficacy. Control assessments are performed at the beginning of the study and at the end of the prospective baseline phase, if applicable and after 4, 8, 12, and 16 weeks. At the end of the first, second, and third treatment week, and at the end of week six, the patient is additionally contacted by telephone. Efficacy and safety parameters are assessed at baseline, during all control visits, and at the end of the study.

ELIGIBILITY:
Inclusion criteria at screening:

* Adult aged between 18 years and 74 years
* Focal epileptic seizures with or without secondary generalization
* Present treatment with one or two antiepileptic drugs (constant dosage during 8 weeks baseline phase prior to initiation of treatment with zonisamide). Stimulation of the vagus nerve is permitted and will not be counted as antiepileptic drug.
* For women of childbearing potential (postmenopausal for more than 1 year): possible pregnancy during the study can be excluded (by hysterectomy, sterilization or simultaneous application of two recognized methods of contraception (no oral contraceptives only)
* For male patients with partners of childbearing potential: a safe method of contraception is practiced during their study participation
* Written consent to participate in the study

Inclusion criteria for randomisation:

* At least 6 focal or clonicotonic seizures documented completely in a seizure diary or the patient chart during the 8 prospective or retrospective weeks baseline phase.

Exclusion criteria at screening:

* Epileptic state during the past year
* Non-epileptic fits
* Generalized epilepsy
* More than 4 weeks of seizure freedom during baseline phase
* Concomitant progressive CNS disease including progressive myoclonus epilepsy
* Concomitant treatment with vigabatrine and / or topiramate
* Hepatic and/or renal insufficiency (creatine > 2mg% or GPT > 2 times ULN)
* Body weight ≤ 40 kg
* (History of) kidney stones; erythrocyturia, family history (in parents, children, brothers and sisters or grandparents) of kidney stones
* (History of) drug and/or alcohol dependence
* Active psychosis
* Suicide attempt during the past 3 years
* Pre-treatment with zonisamide
* Known hypersensitivity to sulfonamides
* concomitant treatment with neuroleptic drugs
* pregnant or breast feeding woman
* participation in another therapy study within 3 months prior to or during this study
* blood donation planned during or within 4 weeks after the participation in this study
* elective surgery planned during the participation in this study
* patient is not willing or not capable to meet the study demands
* patient does not agree to the forwarding of his/her pseudonymous data
* patient without legal competence

Exclusion criteria for randomisation:

- More than 4 consecutive weeks of freedom from seizure during baseline phase

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2005-05; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Change in number of epileptic seizures between week 13 and 16 after start of treatment compared to the correspondently normalized base-line phase. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Christian Elger, Principal Investigator — Universitatsklinikum Bonn, Klinik fur Epileptologie
Locations (30):
- Germany (30):
  - Epilepsieklinik Tabor, Bernau bei Berlin, Brandenburg
  - Universtitatsklinikum Bonn, Bonn, Nordrhein-Westphalen
  - Universtitatsklinikum Munster, Klinik und Poliklinik fur Neurologie, Münster, Nordrhein-Westphalen
  - Epilepsiezentrum Bethel/KSE, Beilefeld
  - Institut fur Diagnostik der Epilepsien Gmbh, Berlin
  - Charite Campus Virchow-Klinikum, Neurologische Klinik und Poliklinik, Berlin
  - St. Josephs Hospital, Neurologische Klinik, Bochum
  - Dr. Gunther Schumann, Bochum
  - Knappschaftskrankenhaus Bochum-Langendreer, Neurologische Klinik, Bochum
  - Dr. Hans Martin Kolbinger, Bonn
  - Neuro-Consil Gmbh, Düsseldorf
  - Neurologische Klinik der Universitat Erlangen, Erlangen
  - Universitatsklinik Essen, Klinik und Poliklinik fur Neurologie, Essen
  - Universitatsklinikum Freiburg, Neurozentrum, Freiburg im Breisgau
  - Universitatsklinikum Gottingen, Abt. fur klinische Neurophysiologie, Göttingen
  - Gemeinschaftpraxis fur Neurologie und Psychiatrie, Hamburg
  - Dr. Heinrich C. Braeuer, Hamburg
  - Ev. Krankenhaus Alsterdorf, Epilepsiezentrum Alsterdorf, Hamburg
  - Epilepsiezentrum Kork, Kehl
  - Epilepsiezentrum Kleinwachau, Epilepsieambulanz, Liegau-Augustusbad
  - Universitatsklinikum Mannheim, Neurologische Klinik, Ambulanz fur Anfallserkrankte, Mannheim
  - Universitatsklinikum, Interdisziplinares Epilepsiezentrum, Marburg
  - Klinikum Grosshadern, Neurologische Klinik und Poliklinik, Epilepsie-Ambulanz, München
  - Klinikum Offenbach, Neurologie, Offenbach
  - Klinik Ernst von Bergmann, Potsdam
  - Universitat Regensburg, Klinik un Poliklinik fur Neurologie, Regensburg
  - Klinik "Die Weissenau", Anfallsambulanz, Revensburg
  - Universitat Rostock, Klinik fur Neurologie und Poliklinik, Rostock
  - Universitatsklinik Ulm Poliklinik fur Neurologie, Epilepsieambulanz, Ulm
  - Dr. Horst-Schmidt Klinik, Neurologie, Wiesbaden